CLINICAL TRIAL: NCT07163949
Title: Balance In Children With Autism Spectrum Disorder: The Role Of Foot Posture And Anthropometry
Brief Title: Balance And Foot Posture In Children With Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Güllü Aydın Yağcıoğlu, Asst Prof, Gulhane School of Medicine
Other Study IDs: AFB
Record Dates: First submitted 2025-08-29; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Autism Disorder; Balance; Posture; Foot Anomalies
Keywords: Autism Spectrum Disorder; Balance; foot; posture; anthropometry
MeSH Terms: conditions — Autistic Disorder; Foot Deformities, Congenital; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Autism Spectrum Disorder: Autism spectrum disorders (ASD) are complex neurodevelopmental conditions characterised by deficits in communication and reciprocal social interactions, as well as restricted interests and repetitive behaviours. Although motor impairments have been recognised as limiting daily motor skills, they are not included in the DSM-5 diagnostic criteria for ASD. The Centers for Disease Control and Prevention published an estimate that the prevalence of ASD in the US population was approximately 1 in 54 eight-year-old children (around 1.85% of the child population). Furthermore, the World Health Organization (WHO) documented a worldwide prevalence of approximately 0.76% in 2010 (affecting nearly 1.16% of the entire child population).
  Interventions: Other: Performance-based tests (such as TUG, foot posture measurements, Tandem Gait test) will be administered to children with ASD.

INTERVENTIONS:
Other: Performance-based tests (such as TUG, foot posture measurements, Tandem Gait test) will be administered to children with ASD. — Children with ASD underwent balance and foot measurement tests that they could perform only by following instructions.

SUMMARY:
The position of the ankle and foot is known as foot posture, and this can have an impact on balance and mobility. Previous research has shown that differences in foot structure and posture between different populations can have a significant impact on balance. However, to our knowledge, no study has examined the relationship between foot posture, anthropometry, muscle strength, and balance in children with Autism Spectrum Disorder. This study was therefore designed to analyse these relationships.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5-18.
* Clinical diagnosis of ASD.

Exclusion Criteria:

* Lack of parental consent;
* Use of assistive devices;
* Presence of vision or hearing loss;
* Use of medications known to impair motor function, such as antipsychotics, stimulants or anticonvulsants;
* Having undergone any lower extremity injury or surgery in the past six months;
* Not being able to follow the commands necessary to obtain the study data.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study included individuals aged 5-18 with a diagnosis of Autism Spectrum Disorder
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Foot Posture Assessment | Baseline
  Foot Posture Assessment: Children's foot posture will be assessed using the Foot Posture Index (FPI-6), which is valid for pediatric individuals. The Foot Posture Index is a scale consisting of a total of 6 items related to the posture of the rear foot and forefoot. These items are talar head palpation, the position of the inclinations above and below the lateral malleolus, the position of the calcaneus, ballooning in the talonavicular joint region, the structure of the medial longitudinal arch, and the abduction/adduction of the forefoot relative to the rearfoot. The total score in this assessment tool ranges from -12 to 12.
Timed Up and Go (TUG) test | Baseline
  Timed Up and Go (TUG) test: For this test, individuals are seated in a chair. The individual is asked to stand up from the chair without assistance, walk three meters on the marked floor, walk back to the chair, and sit down again. The stopwatch is started with the "start" command and stopped when the individual sits down. The TUG time is recorded in seconds (s).
One-Leg Standing Test | Baseline
  One-Leg Standing Test: During this test, which is used to assess an individual's static balance, the subject will be asked to lift one leg without touching the supporting leg, keeping their eyes open, and the time spent on one leg will be recorded in seconds.

SECONDARY OUTCOMES:
Foot-Ankle Anthropometric Measurements | Baseline
  Foot-Ankle Anthropometric Measurements: For the foot-ankle anthropometry of patients, foot length (cm), metatarsal width (cm), and navicular drop height (cm) will be assessed with and without body weight applied to the foot.
Foot Muscle Strength | Baseline
  Foot Muscle Strength: Foot plantar flexion and dorsiflexion muscle strength will be assessed using a digital hand dynamometer.
Tandem Walking Test | Baseline
  Tandem Walking Test: The tandem walking test is used to assess dynamic balance. The subject will be asked to walk along a line drawn on the floor, with the heel of one foot touching the toe of the other foot. The duration of the tandem walk will be measured for each walk, consisting of 10 steps. If balance is lost and the participant is unable to complete 10 steps, the number of steps taken and the duration will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fournier KA, Kimberg CI, Radonovich KJ, Tillman MD, Chow JW, Lewis MH, Bodfish JW, Hass CJ. Decreased static and dynamic postural control in children with autism spectrum disorders. Gait Posture. 2010 May;32(1):6-9. doi: 10.1016/j.gaitpost.2010.02.007. Epub 2010 Apr 18. PMID 20400311
- [Result] Lord C, Elsabbagh M, Baird G, Veenstra-Vanderweele J. Autism spectrum disorder. Lancet. 2018 Aug 11;392(10146):508-520. doi: 10.1016/S0140-6736(18)31129-2. Epub 2018 Aug 2. PMID 30078460